CLINICAL TRIAL: NCT06428006
Title: Efficacy of Cognitive Behavioral Therapy for Insomnia to Treat Insomnia Symptoms and Fatigue in Individuals With Multiple Sclerosis
Brief Title: Efficacy of Cognitive Behavioral Therapy for Insomnia to Treat Insomnia Symptoms in Individuals With Multiple Sclerosis
Acronym: CALM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Catherine Siengsukon, PT, PhD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00160476
Record Dates: First submitted 2024-05-13; First posted 2024-05-24 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Insomnia
Keywords: Cognitive behavioral therapy for insomnia; CBT-I
MeSH Terms: conditions — Multiple Sclerosis; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy for insomnia (Experimental): 1x/week, 6-week 45-60 min one-one-one manualized program via video conferencing (HIPAA-compliant Zoom) with a trained research assistant that includes time in bed restriction, stimulus control, relaxation strategies, cognitive restructuring, and sleep health promotion education.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Sleep and lifestyle education (Active Comparator): 1x/week, 6 weekly 45-60 min one-on-one program via video conferencing (HIPAA-compliant Zoom) with a trained research assistant that includes gentle stretching activities for major muscle groups accompanied by sleep and lifestyle education.
  Interventions: Behavioral: Sleep and lifestyle education

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — The general sessions outlines are as follows with each session:
  Session 1: determine treatment plan, set up sleep schedule and stimulus control, discuss strategies for how to stay awake to prescribed hour and what to do if wake up in middle of night, sleep hygiene education Session 2: continue upward titration of total sleep time, review sleep hygiene; introduce diaphragmatic breathing Session 3: continue upward titration of total sleep time, introduce mindfulness Session 4: continue upward titration of total sleep time, introduce progressive muscle relaxation Session 5: continue upward titration of total sleep time, discuss negative sleep beliefs Session 6: assess global treatment gains, discuss relapse prevention
  Arms: Cognitive behavioral therapy for insomnia
Behavioral: Sleep and lifestyle education — The general sessions outlines are as follows with each session:
  Session 1: Basic sleep education, stretching exercises Session 2: Sleep hygiene education (environmental factors & sleep positions), stretching exercises Session 3: Sleep hygiene education (lifestyle factors), stretching exercises Session 4: Diet recommendations, stretching exercises Session 5: Exercises recommendations, stretching exercises Session 6: Discus maintaining achievements & preventing relapses, stretching exercises
  Arms: Sleep and lifestyle education

SUMMARY:
The incidence of insomnia is estimated to be as high as 90% in individuals with MS due to insomnia being underdiagnosed. Sleep disturbances in people with MS have been associated with reduced cognitive performance, physical function, psychological well-being, quality of life, and occupational function, as well as increased prevalence of fatigue, pain, depression, and anxiety. The objective of the proposed study is to determine the efficacy of cognitive behavioral therapy for insomnia (CBT-I) to improve insomnia symptoms (Aim 1) fatigue, and health-related quality of life (Aim 2) in individuals with multiple sclerosis compared to an active control group, and to determine the characteristics of participants that predict improvement in sleep outcomes (Exploratory Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosis of relapsing-remitting or secondary progressive MS based on established guidelines20 and verified by their neurologist
* Mild-to-moderately severe disability (≤ 6 on Patient Determined Disability Steps (PDDS) scale)
* Report of difficulty falling asleep, maintaining sleep, or waking up too early at least 3 nights/week for the past 3 months with significant distress and impact on function despite adequate opportunity for sleep and not due to other sleep disorders as indicated in the DSM-5
* ≥10 on Insomnia Severity Index
* English speaking
* ≥31 on modified Telephone Interview of Cognitive Status23
* Has a high school diploma or equivalent to serve as a proxy measurement of reading ability to ensure adequate reading ability to participate in the study
* Report having access to internet service or a data plan and access to a computer, tablet, or smart phone

Exclusion Criteria:

* Known untreated sleep disorder (such as sleep apnea or restless legs syndrome)
* >3 on STOP BANG indicating increased risk of sleep apnea
* Restless legs syndrome as determined by RLS-Diagnosis Index
* Circadian rhythm sleep-wake disorder as determined by the Sleep Disorders-Revised
* Parasomnia as determined by the Sleep Disorders-Revised
* Currently taking benzodiazepines, non-benzodiazepines, or melatonin supplements or agonists for insomnia
* Score of ≥20 on the Patient Health Questionnaire (PHQ-9) indicating severe depression or endorsement of suicidal ideation (answer 1, 2 or 3 on #9 of the PHQ-9)
* Score of ≥15 on the Generalized Anxiety Disorder (GAD-7) indicating severe anxiety
* Current or history (up to 2 years) of alcohol or drug or alcohol abuse as indicated by DSM-5 criteria
* History of other nervous system disorder such as stroke or Parkinson's disease
* Currently pregnant or intending to become pregnant in the next 6 months
* Severe mental illness such as schizophrenia or bipolar disorder
* Severe neurological or sensory impairments that would interfere significantly with testing
* Relapse and/or corticosteroid use in the past 8 weeks
* History of (within 5 years) or currently conducting overnight shift work including hours of midnight-4am
* Currently receiving a behavioral sleep health intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | baseline, Week 6, Month 6
  The ISI consists of 7 questions, each rated on a 0-4 scale. The range of scores on the ISI is 0-28, with a score of ≥ 10 suggesting clinical insomnia. The lower the score the less severe insomnia.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | baseline, Week 6, Month 6
  The PSQI consists of 9 items within 7 sleep categories. The 7 sleep category scores are summed to form a single global score ranging from 0-21. A global score of >5 reflects poor sleep quality.
Epworth Sleepiness Scale (ESS) | baseline, Week 6, Month 6
  Consists of eight scenarios of daily activity, and participants use a four-point Likert scale to rate how likely they are to doze. Score ranges 0-24 with a higher score indicating daytime sleepiness.
Dysfunctional Beliefs About Sleep | baseline, Week 6, Month 6
  This assessment is a 10 item Likert-scale self-report questionnaire. Higher scores indicate more dysfunctional beliefs.
Positive Affect and Negative Affect Schedule (PANAS) | baseline, Week 6, Month 6
  is a 20-item self-report questionnaire used to measure positive and negative emotions. There are two subscales (Positive Affect and Negative Affect) with 10 items each. The respondent scores how applicable a list of emotions are on a 5-point Likert scale with 1 = "Very slightly or not at all" to 5 = "Extremely". A higher score on the Positive Affect subscale indicates greater intensity of positive emotions, and a high score on Negative Affect indicate greater intensity of negative emotions.
Sleep Self-Efficacy Scale (SESS) | baseline, Week 6, Month 6
  Sleep Self-Efficacy is a 9 item self-report Likert-scale questionnaire use to identify sleep self-efficacy. Scores range from 0-45 and a higher score indicates higher sleep self-efficacy.
Actigraphy | baseline, Week 6, Month 6
  Participants will wear an actigraph on their non-dominant wrist for 7 nights to assess sleep/wake cycle. Mains variables of interest are sleep regularity, timing, efficiency, and duration
Modified Fatigue Impact Scale (MFIS) | baseline, Week 6, Month 6
  The MFIS assesses the impact of fatigue on daily activities for the month prior. The MFIS consists of 21 items with 3 subscales: physical, cognitive, and psychosocial. The score on the 21 items are scored with a range of 0-84 with a higher score indicating a greater impact of fatigue.
Fatigue Severity Scale (FSS) | baseline, Week 6, Month 6
  The FSS assesses the impact of fatigue on activities for the week prior and consists of 9 questions. The mean of the 9 scores is calculated with a range of 0-7.
Multiple Sclerosis Impact Scale (MSIS-29) | baseline, Week 6, Month 6
  Quality of life will be assessed using the Multiple Sclerosis Impact Scale (MSIS-29). MSIS-29 is total of 29 items scale, with subscales of physical (20 items) and psychological (9 items). Responses computed in a range from 0-100, and higher scores indicating a worse quality of life due to physical and physiological impacts of MS
Cognitive Failures Questionnaire (CFQ) | baseline, Week 6, Month 6
  Cognitive Failures Questionnaire (CFQ) assesses perception of cognitive abilities over the past 6 months. consists of 25 items that the individual rates on a 5-point Likert scale with 0 = "never" and 4 = "Very Often" with a summary score of 0-100 with a higher score indicating poorer perceived cognitive abilities.

OTHER OUTCOMES:
Patient-Determined Disability Steps (PDDS) | baseline
  Disability will be assessed using the PDDS scale which is a single-item 9 point scale ranging from "normal" (score of 0) to "bedridden" (score of 8).
Patient Health Questionnaire (PHQ-9) | baseline, Week 6, Month 6
  Depressive symptoms will be assessed using the 9-item Patient Health Questionnaire (PHQ-9), with a score of ≥20 suggesting severe depression. It consists of 9 items with a score ranging from 0-27.
Generalized Anxiety Disorder Assessment (GAD-7) | baseline, Week 6, Month 6
  Anxiety symptoms will be assessed using the 7-item GAD-7, with a score of ≥15 indicating severe anxiety. This questionnaire consists of 7 items, and the score from each item is summed for an overall score ranging from 0-21 with a higher score indicating a higher level of anxiety
Adherence to CBT-I intervention | Each CBT-I session Week 1-6
  To assess adherence to the CBT-I intervention, the sleep log will be used to assess number of mornings/week got out of bed at agreed upon time and the number of times got out of bed if unable to sleep. A total percentage will be calculated and used as the outcome of interest.
Diet quality | baseline
  Participants will be asked "In general, how healthy is your overall diet?" and will rate on a 5-point Likert scale (5 = "excellent", 4 = "very good", 3 = "good", 2 = "fair", 1 = "poor")
Eating regularity | baseline, Week 6, Month 6
  Participants will mark on the sleep log at each assessment period the time period for eating breakfast, lunch, and dinner. Variability in mealtime will be quantified as the standard deviation from the individual's mean meal start time.
Nighttime urination frequency | baseline, Week 6, Month 6
  Participants will mark on the sleep log the number of times they wake up to void their bladder during the sleep opportunity window.
PainDetect | baseline, Week 6, Month 6
  PainDetect includes 13 items that assesses neuropathic pain. A total score ranges from -1 to 38, with higher scores indicating higher levels of neuropathic pain.
Fibromyalgia Survey Questionnaire | baseline, Week 6, Month 6
  Fibromyalgia Survey Questionnaire includes the assessment of the number of painful body regions. Scores ranges from 0-31. A higher score indicates worse symptoms.
PROMIS SF v.1.0 - Pain Intensity | baseline, Week 6, Month 6
  Measures max and average pain intensity during past 7 days. The T-score value, with a mean of 50 and standard deviation of 10 representing the rescaled raw score, will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siengsukon CF, Robichaud J, Nelson E, Glaser A, Baber GR, Gratton MKP, Zanotto A, Phadnis MA, Lynch S. Cognitive behavioral therapy for insomnia for individuals with multiple sclerosis (CALM): A randomized control trial protocol. Contemp Clin Trials Commun. 2026 Jan 10;49:101595. doi: 10.1016/j.conctc.2026.101595. eCollection 2026 Feb. PMID 41626064